CLINICAL TRIAL: NCT05578612
Title: Timing of Bridge Plate Removal and Distal Radius Fracture Outcomes: A Multicenter Randomized, Controlled Trial
Brief Title: Timing of Bridge Plate Removal and Distal Radius Fracture Outcomes
Acronym: TORPEDO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn following PI departure from Sponsor institution.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01142
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Distal Radius Fracture
Keywords: Fracture of Lower End of Radius
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridge Plate Removal at 6-8 Weeks Postoperatively (Experimental): Participants will undergo dorsal spanning bridge plate fixation per standard technique. Patients in the experimental group will return to the operative room for removal of the bridge plate at Week 6-8. Patients will begin the standardized postoperative rehabilitation protocol immediately following bridge plate removal on Week 6-8.
  Interventions: Procedure: Dorsal Spanning Bridge Plate Fixation; Procedure: Dorsal Spanning Bridge Plate Removal
- Bridge Plate Removal at 12-14 Weeks Postoperatively (Active Comparator): Participants will undergo dorsal spanning bridge plate fixation per standard technique. Patients in the control group will return to the operating room for removal of the bridge plate at Week 12-14. Patients will begin the standardized postoperative rehabilitation protocol immediately following bridge plate removal on Week 12-14.
  Interventions: Procedure: Dorsal Spanning Bridge Plate Fixation; Procedure: Dorsal Spanning Bridge Plate Removal

INTERVENTIONS:
Procedure: Dorsal Spanning Bridge Plate Fixation — Dorsal spanning bridge fixation will be performed by board-certified orthopedic surgeons per standard technique.
Procedure: Dorsal Spanning Bridge Plate Removal — Dorsal spanning bridge removal will be performed by board-certified orthopedic surgeons per standard technique.

SUMMARY:
The purpose of this randomized control trial will be to determine whether the duration of bridge plate fixation of distal radius fractures can be reduced to 6-8 weeks without worsening of functional outcomes relative to the current standard of greater than 12 weeks of fixation. The secondary aim of the study is to determine whether a reduced duration of bridge plate fixation leads to an increase in wrist range of motion following plate removal compared to the standard duration of fixation. 100 patients with comminuted distal radius fractures that are indicated for bridge plate fixation will be randomized to the Accelerated Removal arm (n = 50) or the Standard Removal arm (n = 50).

ELIGIBILITY:
Inclusion Criteria:

1. Fracture of the distal radius indicated for operative treatment using bridge plate fixation
2. Age 18 years or greater
3. Capacity to provide informed consent

Exclusion Criteria:

1. Bridge plate fixation in the setting of revision surgery for prior nonunion or malunion
2. Bilateral distal radius fractures (prevents accurate measurement of postoperative range of motion and strength of the injured extremity without a normal contralateral extremity for comparison)
3. Pathologic fractures
4. Patients that will be unable to complete the necessary follow up, including incarcerated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Disabilities of the Arm, Shoulder, and Hand (DASH) Score | Baseline, Week 104
  30-item questionnaire that asks the patient to rate their difficulty with common functional tasks and the severity of upper extremity symptoms over the past week. DASH is reported on a scale of 0-100 with lower scores indicating less severe symptoms and superior function. A decrease in scores indicates symptoms became less severe and function improved during the observational period.

SECONDARY OUTCOMES:
Change in Patient-Related Wrist Evaluation (PRWE) Questionnaire Score | Baseline, Week 104
  15-item questionnaire related to wrist pain and function during typical activities of daily living. Items are rated on a Likert scale from 0 (no pain or difficulty) to 10 (the worst pain you have ever experienced or you could not do the task). The total score ranges from 0-100; higher scores indicate greater disability. An increase in scores indicates disability increased during the observational period.
Change in Volar Tilt | Removal of Bridge Plate (from Week 6 to up to Week 14), Week 104
  Approximation of displacement in the sagittal plane. Radiographs taken immediately after bridge plate removal will be compared to final radiographs at the conclusion of the study period.
Change in Radial Inclination | Removal of Bridge Plate (from Week 6 to up to Week 14), Week 104
  Approximation of displacement in the coronal plane. Radiographs taken immediately after bridge plate removal will be compared to final radiographs at the conclusion of the study period.
Change in Radial Height | Removal of Bridge Plate (from Week 6 to up to Week 14), Week 104
  Approximation of displacement in the coronal plane. Radiographs taken immediately after bridge plate removal will be compared to final radiographs at the conclusion of the study period.
Change in Ulnar Variance | Removal of Bridge Plate (from Week 6 to up to Week 14), Week 104
  Approximation of displacement in the coronal plane. Radiographs taken immediately after bridge plate removal will be compared to final radiographs at the conclusion of the study period.
Range of Motion: Flexion-Extension Arc Relative to Contralateral Side | Up to Week 104
  Range of Motion (ROM) will be measured using a digital goniometer. The ROM of the operative extremity will be expressed as a percentage of the operative wrist ROM relative to the uninjured wrist ROM. The arc of motion will be measured 3 times per visit and averaged for both the operative extremity and the contralateral extremity.
Range of Motion: Pronosupination Arc Relative to Contralateral Side | Up to Week 104
  Range of Motion (ROM) will be measured using a digital goniometer. The ROM of the operative extremity will be expressed as a percentage of the operative wrist ROM relative to the uninjured wrist ROM. The arc of motion will be measured 3 times per visit and averaged for both the operative extremity and the contralateral extremity.
Range of Motion: Ulnar-Radial Deviation Arc Relative to Contralateral Side | Up to Week 104
  Range of Motion (ROM) will be measured using a digital goniometer. The ROM of the operative extremity will be expressed as a percentage of the operative wrist ROM relative to the uninjured wrist ROM. The arc of motion will be measured 3 times per visit and averaged for both the operative extremity and the contralateral extremity.
Isometric Force: Grip Force Relative to Contralateral Side | Up to Week 104
  Isometric force will be measured using a handheld dynamometer. Force measurements will be repeated 3 times per visit in both extremities. The force produced by the operative extremity will be expressed as a percentage of the operative wrist force relative to the uninjured wrist force.
Isometric Force: Wrist Extension Force Relative to Contralateral Side | Up to Week 104
  Isometric force will be measured using a handheld dynamometer. Force measurements will be repeated 3 times per visit in both extremities. The force produced by the operative extremity will be expressed as a percentage of the operative wrist force relative to the uninjured wrist force.
Isometric Force: Wrist Flexion Force Relative to Contralateral Side | Up to Week 104
  Isometric force will be measured using a handheld dynamometer. Force measurements will be repeated 3 times per visit in both extremities. The force produced by the operative extremity will be expressed as a percentage of the operative wrist force relative to the uninjured wrist force.
Incidence of Nonunion at Surgical Site | Up to Week 104
  Nonunions will be defined based on the presence of both clinical and radiographic evidence of failed bony union after 8 weeks as agreed upon by two independent orthopedic surgeons. Pain, tenderness, and detectible motion at the fracture site will serve as clinical indicators of nonunion. Lack of bridging callus at the fracture site on plain radiographs taken coplanar with the fracture will serve as direct evidence of nonunion.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Azad, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Ali.Azad@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Ali.Azad@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.